CLINICAL TRIAL: NCT07189468
Title: AI-based Progression and Medication Response Prediction Study in Parkinson's Disease
Acronym: AI-PMP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Aristotle Univ. of Thessaloniki (Greece) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC31/25/0193
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: AI; Parkinson disease; smartwatch
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Polygenic risk score
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Parkinson's disease patients: Parkinson's disease patients to be monitored via a smartwatch and a mobile application
  Interventions: Device: Smartwatch and mobile application

INTERVENTIONS:
Device: Smartwatch and mobile application — Wearing a smartwatch and using a mobile application for one year

SUMMARY:
The study aims to provide initial PoC validation data of two AI models to predict disease progression and treatment side effects in PD patients using as input patients' demographic, clinical and genetic information, as well as digital biomarker measurements in daily living collected via a smartwatch and a mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease diagnosis according to MDS criteria (Postuma et al., 2015)
* Disease duration ranging from 5 to 10 years
* Age 40-80
* Patients in stages 2 and 3 of the Hoehn and Yahr (a functional disability scale) in the ON condition
* The participant is using a compatible smartphone
* Written informed consent

Exclusion Criteria:

* Atypical Parkinsonian Syndrome
* Second-line device-aided treatments
* Patients with >4 daily doses of L-DOPA
* Daily levodopa equivalent dose > 1500 mg
* Ongoing hallucinations requiring short-term treatment adjustment
* Inability to provide informed consent or participate in the study
* Inability to use the smartwatch and/or the mAI-Care app - as judged by investigator
* Lacking motivation to participate in study procedures - as judged by investigator
* Under adult autonomy protection system, legal guardianship or incapacitation
* Pregnant and breast-feeding women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Classification performance of the Parkinson's disease (PD) progression prediction model | Between baseline and 12 months
  Classification performance of the model in predicting observed motor disease progression, defined as a binary outcome: the condition of a patient is classified as worsened if either the Movement Disorder Society Unified Parkinson's Disease (MDS-UPDRS) rating scale part III score in ON-state increases by more than 3 points (>3), or the Levodopa Equivalent Daily Dose (LEDD) increases by more than 10%.

SECONDARY OUTCOMES:
Usability of the mAI-Care app | 12 month visit
  System Usability Scale score of end-users (PD patients)
Usability of the mAI-Insights app | 12 month visit
  System Usability Scale score of end-users (clinicians)

CONTACTS AND LOCATIONS:
Locations (4):
- University Hospital of Toulouse, Toulouse, France
- Technische Universität Dresden, Dresden, Germany
- Hospital Ruber Internacional, Madrid, Spain
- Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No